CLINICAL TRIAL: NCT01167985
Title: Clinical Study: Evaluation of the Antibacterial Effect of Insoluble Antibacterial Nanonparticles Incorporated in Dental Materials for Endodontic Treatment
Brief Title: A Clinical Study: the Antibacterial Effect of Insoluble Antibacterial Nanoparticles (IABN) Incorporated in Dental Materials for Root Canal Treatment
Acronym: IABN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Perez Davidi Michael, DMD, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191062 HMO-CTIL
Record Dates: First submitted 2010-06-09; First posted 2010-07-22 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Endodontic Treatment; Irreversible Pulpitis; Health Pulp; Infected Pulp
Keywords: antibacterial polyethyleneimine nanoparticles; quaternary ammonium; dental; Endodotnic; pulp; bacteria; Root canal sealer; temporary filling; provisional restoration

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Root canal sealer group+ IABN (Experimental): Device: alkylated polyethylenimine nanoparticles antibacterial evaluation
  Interventions: Device: IABN
- Provisional restoration material+ IABN (Experimental): Device: alkylated polyethylenimine nanoparticles antibacterial evaluation
  Interventions: Device: IABN
- Experimental- Different root canal sealer+ IABN (Experimental): Device: alkylated polyethylenimine nanoparticles antibacterial evaluation
  Interventions: Device: IABN

INTERVENTIONS:
Device: IABN — Patients with single canal teeth diagnosed with infected pulp and periapical lesion, and need root canal treatment, will be asked to participate in the study. The study group will have their canal sealed with endodontic sealer + the nanoparticles. The control group will have their canal sealed with the conventional sealer alone. The patients will be invited to 4 follow ups during which a clinical and radiological examinations will be performed.While preparing the post, a sample of the sealer will be taken to evaluation in the lab.
  Other Names: QA-PEI
  Arms: Root canal sealer group+ IABN
Device: IABN — patients with molar teeth diagnosed with healthy pulp or irreversible pulpitis, and need root canal treatment, will be asked to participate in the study. After cleaning the teeth following a standard protocol, a sterile cotton wool will be placed in the pulp chamber. provisional restoration with and without nanoparticles will seal the teeth between apointments. After a month the cotton wool will be taken out and tansferred to the laboratory. The root canal treatment will continue following the standard protocol.
  Other Names: QA-PEI
  Arms: Provisional restoration material+ IABN
Device: IABN — Patients with single canal teeth diagnosed with infected pulp and periapical lesion, and need root canal treatment, will be asked to participate in the study. The study group will have their canal sealed with endodontic sealer + the nanoparticles. The control group will have their canal sealed with the conventional sealer alone. The patients will be invited to 4 follow ups during which a clinical and radiological examinations will be performed.While preparing the post, a sample of the sealer will be taken to evaluation in the lab.
  Other Names: QA-PEI
  Arms: Experimental- Different root canal sealer+ IABN

SUMMARY:
The effect of Antibacterial Nanoparticles, Incorporated in root canal sealer material and in provisional restoration is going to be examined. Two different tests are planned: (1) clinical and radiological evaluation of root canal sealer.(2) An evaluation in the laboratory the efficacy of provisional restoration during root canal treatment.We assume, based on our previous laboratory studies that show antibacterial properties, that the incorporation of the nanoparticels will improve the treatment outcome.

DETAILED DESCRIPTION:
1. patients with molar teeth diagnosed with healthy pulp or irreversible pulpitis, and need root canal treatment, will be asked to participate in the study. After cleaning the teeth following a standard protocol, a sterile cotton wool will be placed in the pulp chamber. provisional restoration with (test group-40 patients) and without (control group- 40 patients) nanoparticles will seal the teeth between apointments. After a month the cotton wool will be taken out and tansferred to the laboratory. The root canal treatment will continue following the standard protocol.
2. patients with single canal teeth diagnosed with infected pulp and periapical lesion, and need root canal treatment, will be asked to participate in the study. Two study group (40 patients on each group) will have their canal sealed with a two types of endodontic sealers each + the nanoparticles. The control group (40 patients) will have their canal sealed with the conventional sealer alone. The patients will be invited to 4 follow ups: 2 weeks, 3 months, 6 months and 1 year during which a clinical and radiological examinations will be performed.While preparing the post, a small example of the sealer will be taken to a test in the lab.

ELIGIBILITY:
Inclusion Criteria:

1. Needs root canal treatment
2. For the provisional restoration- molar teeth with class II restoration
3. For the provisional restoration-healty/ uninfected teeth
4. For the root canal sealer- single root canal
5. For root canal sealer-infected teeth

Exclusion Criteria:

1. systemic health problems
2. Pregnant women
3. The use of antiseptic mouth rinse or antibiotic Up to 2 weeks before the beginning of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
In vitro evaluation | One month for provisional restoration.
  clinical and radiological evaluation of the radiolucent periapical lesion, for the root canal sealer. As for the provisional restoration, in vitro assesment of bacterial growth.

SECONDARY OUTCOMES:
Radiological evaluation of the root canal sealer | 1 year for the root canal sealer.
  clinical and radiological evaluation of the radiolucent periapical lesion, for the root canal sealer. As for the provisional restoration, in vitro assesment of bacterial growth.
Clinical and in vitro evaluation of the root canal sealer | 1 year for the root canal sealer.
  clinical and radiological evaluation of the radiolucent periapical lesion, for the root canal sealer. As for the provisional restoration, in vitro assesment of bacterial growth.While preparing the post, a sample of the sealer will be taken to evaluation in the lab.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Michael Perez Davidi, DMD, Principal Investigator — Hadassah Medical Organization; Ervin Weiss, DMD, Study Chair — Hadassah Medical Organization; Itzhak Abramovitz, DMD, Study Chair — Hadassah Medical Organization; Dana Kesler Shvero, DMD, Study Chair — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Beyth N, Yudovin-Farber I, Bahir R, Domb AJ, Weiss EI. Antibacterial activity of dental composites containing quaternary ammonium polyethylenimine nanoparticles against Streptococcus mutans. Biomaterials. 2006 Jul;27(21):3995-4002. doi: 10.1016/j.biomaterials.2006.03.003. Epub 2006 Mar 27. PMID 16564083
- [Background] Slutsky H, Weiss EI, Lewinstein I, Slutzky S, Matalon S. Surface antibacterial properties of resin and resin-modified dental cements. Quintessence Int. 2007 Jan;38(1):55-61. PMID 17216909
- [Background] Matalon S, Weiss EI, Gozaly N, Slutzky H. Surface antibacterial properties of compomers. Eur Arch Paediatr Dent. 2006 Sep;7(3):136-41. doi: 10.1007/BF03262554. PMID 17140542
- [Background] Yudovin-Farber I, Beyth N, Nyska A, Weiss EI, Golenser J, Domb AJ. Surface characterization and biocompatibility of restorative resin containing nanoparticles. Biomacromolecules. 2008 Nov;9(11):3044-50. doi: 10.1021/bm8004897. Epub 2008 Sep 27. PMID 18821794
- [Background] Shvero DK, Davidi MP, Weiss EI, Srerer N, Beyth N. Antibacterial effect of polyethyleneimine nanoparticles incorporated in provisional cements against Streptococcus mutans. J Biomed Mater Res B Appl Biomater. 2010 Aug;94(2):367-371. doi: 10.1002/jbm.b.31662. PMID 20583306
- See also: Michael Perez Davidi — http://www.mypd.co.il